CLINICAL TRIAL: NCT07120750
Title: The Impact of Different Antiviral Strategies on Tumor Prognosis in Patients With HBV-related Liver Cancer After Radical Treatment: A Prospective, Open-label, Non-randomized Clinical Study
Brief Title: Post-Radical Treatment Antiviral Strategies in HBV-Related Liver Cancer: Impact on Tumor Prognosis
Acronym: PRTRAS 001
Status: Not yet recruiting | Type: Observational
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2024-077
Record Dates: First submitted 2025-07-08; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC); Chronic Hepatitis B
Keywords: Hepatocellular carcinoma; Peginterferon alfa-2b; Nucleos(t)ide analogues; Post-radical treatment; Clinical cure
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B, Chronic | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will retain the following biospecimens:
  1. Blood serum samples: Collected at regular intervals to measure HBV DNA levels, HBsAg status, and liver function parameters, and to assess treatment effectiveness and monitor adverse events.
  2. Peripheral blood mononuclear cells (PBMCs): Isolated from blood samples to evaluate immune response to treatment and for future research on host-virus interactions.
  3. Surgically resected liver cancer tissue: Collected for pathological analysis of tumor characteristics and molecular studies on treatment effects and biomarkers linked to recurrence.
  4. Peritumoral liver tissue: Samples from the tissue adjacent to the cancer will be collected to study the tumor microenvironment and compare molecular and pathological features between cancerous and non-cancerous tissue.
  All samples will be anonymized, stored securely, and used for analyses in line with the study's objectives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Intervention for Group 1 — Participants will receive standard NAs therapy, which may include entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide fumarate (TAF), or tenofovir amibufenamide (TMF). NAs are antiviral medications used to suppress HBV replication and manage chronic hepatitis B infection.
Drug: Intervention for Group 2 — Participants will receive Peg-IFNα-2b in addition to NAs therapy. Peg-IFNα-2b is an antiviral medication that works by boosting the immune system and has additional antiviral, antifibrotic, and anti-tumor effects. It is used to treat chronic hepatitis B and may help reduce the recurrence of liver cancer.

SUMMARY:
The goal of this clinical trial is to learn if peginterferon alfa-2b can reduce the recurrence of HBV-related liver cancer in patients who have undergone radical treatment. The study will also explore the potential benefits of peginterferon alfa-2b in achieving clinical cure and its impact on reducing liver cancer recurrence.

The trial is designed as a single-center, non-randomized, open-label study. Participants will be HBV-related liver cancer patients who have received radical treatment. The study will compare two groups: one receiving nucleos(t)ide analogues (NAs) alone and the other receiving NAs combined with peginterferon alfa-2b. The main question it aims to answer is:

Can peginterferon alfa-2b lower the 3-year recurrence rate in HBV-related liver cancer patients after radical treatment?

Participants will undergo regular follow-ups, including imaging studies and blood tests, to monitor for cancer recurrence and assess the safety of the treatment.

DETAILED DESCRIPTION:
1. Study Background The 3-year recurrence rate of HBV-related liver cancer after radical surgery is as high as 40% to 70%. This study aims to explore whether the addition of peginterferon alfa-2b (Peg-IFNα-2b) to nucleoside (acid) analogues (NAs) can reduce the risk of recurrence through immune modulation.
2. Key Mechanism Hypotheses

   Peg-IFNα-2b may reduce the reactivation of micrometastases through:
   * Enhancing HBV-specific T-cell responses
   * Lowering serum HBsAg levels
   * Inhibiting immune suppression in the tumor microenvironment
3. Detection Methods

   * Imaging Monitoring: Abdominal MRI (using LI-RADS v2018 criteria) every 12 weeks ± 7 days.
   * Laboratory Tests:
   * HBV DNA: COBAS® TaqMan HBV Test (LLOQ = 10 IU/mL)
   * Quantitative HBsAg: Architect HBsAg QT assay
   * PBMC Immune Profile: Flow cytometry (proportion of CD8+/PD-1+ T cells)
   * Tissue Biomarkers: Postoperative tumor tissue PD-L1 immunohistochemistry (22C3 antibody) and T-cell infiltration score.
4. Statistical Design

   * Sample size: 332 cases (power 80%, α = 0.05, expected HR = 0.6)
   * Primary endpoint analysis: 3-year cumulative recurrence rate (Kaplan-Meier method + Log-rank test)
   * Covariate adjustment: Cox model includes age, BCLC stage, and baseline HBsAg level.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 18 and 70 years of age.
* HBsAg Positive: Participants must be positive for hepatitis B surface antigen (HBsAg).
* Confirmed Hepatocellular Carcinoma (HCC): Participants must have a pathological confirmation of HCC via surgical resection or local ablation.
* BCLC Staging: Participants must have a Barcelona Clinic Liver Cancer (BCLC) staging of 0 or A.
* Liver Function: Participants must have normal or well-compensated liver function, classified as Child-Pugh A.
* Expected Survival: Participants must have an expected survival of more than 3 months.
* Informed Consent: Participants must sign an informed consent form and agree to comply with the study requirements. If a participant is unable to sign the consent form, a legal guardian or agent must do so.

Exclusion Criteria:

* Prior Systemic Cancer Treatments: Participants who have received prior systemic cancer treatments such as liver transplantation, chemotherapy, targeted therapy, or biological therapy will be excluded.
* Other Active Malignancies: Participants with a history or presence of other active malignancies, except for skin basal cell carcinoma or squamous cell carcinoma that has been cured, or cervical carcinoma in situ, will be excluded.
* Allergies to Interferon: Participants who are allergic to interferon or any of its components, or whom the investigator deems unsuitable for interferon therapy, will be excluded.
* Other Chronic Liver Diseases: Participants with other chronic liver diseases such as hepatitis A, C, D, or E virus infection, alcoholic liver disease, genetic metabolic liver disease, or drug-induced liver disease will be excluded.
* Autoimmune Diseases:Participants with autoimmune diseases,including autoimmune liver disease and psoriasis, will be excluded.
* Severe Liver Dysfunction: Participants with severe liver dysfunction or decompensated cirrhosis will be excluded.
* Renal Impairment: Participants with serum creatinine levels exceeding 1.5 times the upper limit of normal will be excluded.
* Severe Systemic Diseases:Participants with severe systemic diseases affecting the heart,lungs,kidneys,brain,or blood will be excluded.
* Severe Neuropsychiatric Disorders:Participants with severe neuropsychiatric disorders such as epilepsy, depression, mania, or schizophrenia will be excluded.
* Unstable Medical Conditions:Participants with unstable diabetes,hypertension,hyperthyroidism,or other endocrine diseases will be excluded.
* Retinopathy:Participants with a history of severe retinopathy or other evidence of retinopathy will be excluded.
* Substance Abuse:Participants with a history of drug abuse or alcoholism will be excluded.
* Pregnancy or Breastfeeding:Pregnant or breastfeeding women, or women planning to become pregnant during the study period who are unwilling to use contraception, will be excluded.
* Investigator's Judgment:Participants whom the investigator deems unsuitable for the study based on their current medical condition will be excluded.
* Concurrent Participation in Other Trials:Participants who are concurrently involved in other clinical research trials will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adults aged 18 to 70 with HBV-related liver cancer who have undergone radical treatment (surgery or ablation). They are HBsAg-positive, with pathological confirmation of HCC and BCLC staging of 0 or A. Participants must have adequate liver function (Child-Pugh A), an expected survival of over 3 months, and provide informed consent. The study excludes those with prior systemic cancer treatments, other active malignancies, allergies to interferon, severe liver or renal dysfunction, and other significant health issues.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
3-Year Cumulative Recurrence Rate via MRI (LI-RADS) | 3 years post-radical treatment.
  1. Measurement Tool: Liver Imaging Reporting and Data System (LI-RADS v2018) 1.1 Primary modality: Dynamic contrast-enhanced MRI 1.2 Confirmatory criteria: 1.2.1 LI-RADS 5 (definite HCC): 1.2.1.1 Arterial hyperenhancement + 1.2.1.2 Portal venous washout ± 1.2.1.3 Capsule/threshold growth 1.2.2 Histopathology (biopsy) for equivocal cases
  2. Definition: Proportion of participants with new intrahepatic lesions meeting LI-RADS 5 criteria or histologically confirmed HCC metastases within 3 years post-radical treatment.
  3. Clinical Significance: Recurrence defined as:
  3.1 Local (original site) 3.2 Intrahepatic (>2 cm from resection margin) 3.3 Extrahepatic (metastases with biopsy confirmation)

SECONDARY OUTCOMES:
2-Year HBsAg Seroclearance Rate | 2 years post-treatment initiation.
  * Measurement Tool: Architect HBsAg QT Assay
  * Definition: Proportion with HBsAg loss (<0.05 IU/mL)
  * Directionality: Lower HBsAg levels indicate better response
  * Confirmation: Required at two timepoints ≥24 weeks apart
2-Year HBV DNA undetectable rate | 2 years post-treatment initiation.
  * Measurement Tool: COBAS® TaqMan HBV Test v2.0
  * Definition: Proportion of participants achieving HBV DNA <10 IU/mL (LLOQ) in two consecutive tests ≥6 months apart
  * Directionality: Lower values indicate better virological control
Incidence of Adverse Events (AEs) | Throughout the 3-year follow-up period.
  * Measurement Tool: CTCAE v5.0 grading system
  * Definition: Frequency of all-cause AEs, categorized by:
  * Severity: Grade 1 (mild) to 5 (death)
  * Relatedness: Definite/probable/possible vs. unrelated
  * Range: 1-5 scale (higher grade = worse severity)
  * Reporting Threshold: All events ≥Grade 2
Serious Adverse Event (SAE) Rate | Throughout the 3-year follow-up period.
  * Measurement Tool: CTCAE v5.0
  * Definition: Events meeting ≥1 SAE criterion:
  Death/life-threatening Hospitalization/prolonged hospitalization Persistent disability Congenital anomaly
  -Causality Assessment: Using WHO-UMC system
Liver Function Deterioration Rate | Throughout the 3-year follow-up period.
  * Measurement tool: Change in Child-Pugh score ≥ 2 points
  * Range: 5 - 15 points (the higher the score, the worse the liver function)
  * Definition: The proportion of patients with an increase in Child-Pugh score of ≥ 2 points during treatment compared to the baseline.
Quality of Life Change | Throughout the 3-year follow-up period.
  * Measurement tool: EORTC QLQ-C30
  * Range: 0-100 (higher scores on functional dimensions indicate better status; higher scores on symptom dimensions indicate worse status)
  * Definition: Change from baseline in global health status/QoL over 3 years, analyzed with a mixed-effects linear model.

IPD SHARING:
Plan to Share IPD: Yes
1. Data Availability: De-identified individual participant data will be made available upon reasonable request after the completion of the study and publication of the primary results.
  2. Time Frame: Data will be available starting from six months after the publication of the primary study results and for a period of five years thereafter.
  3. Access Criteria:
  (1) Requests for data access will be reviewed by the study's data monitoring committee.
  (2) Data will be shared for research purposes that are consistent with the original study objectives and for the advancement of scientific knowledge.
  (3) Researchers requesting access must submit a detailed proposal outlining their research question, methods, and analysis plan.
  4. Data Sharing Process:
  1. Data will be provided in a de-identified format, ensuring participant confidentiality.
  2. Along with the data, relevant documentation such as the study protocol, statistical analysis plan, and data dictionary will be made available to facili
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: * Start Date: Six months after the publication of the primary study results.
  * End Date: Five years following the start date.
  * Description: "De-identified individual participant data will be available starting six months after the publication of the primary study results and for a period of five years thereafter."
Access Criteria: * Who Can Access: Researchers who submit a valid research proposal outlining a scientific objective that is consistent with the original study aims.
  * What Can Be Accessed: De-identified dataset along with relevant study documentation (e.g., protocol, statistical analysis plan, data dictionary).
  * How to Access: By submitting a formal request to the principal investigator, including a detailed research proposal and data usage plan. Access will be granted upon approval by the study's data monitoring committee.
  * Description: "Access to the de-identified individual participant data and supporting documentation will be granted to qualified researchers upon approval of a formal request and research proposal. Researchers must demonstrate that their objectives align with the original study's scope."
URL: http://www.szsdsrmyy.com/